CLINICAL TRIAL: NCT04962594
Title: Safety and Efficacy of Starter Infant Formula, Follow-up Formula and Growing-up Milk Supplemented With Pre- and Probiotic(s): a Double-blind, Randomized, Controlled Trial
Brief Title: Safety and Efficacy of Infant Formulas Supplemented With Pre- and Probiotic(s)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20.12.INF
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy Infants
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, controlled trial plus a non-randomized breastfed reference group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unique coding of the study products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental formulas (EF) group (Experimental): Starter infant formula, follow-up infant formula and growing-up milk (partially hydrolyzed bovine whey protein) supplemented with pre- and probiotic(s)
  Interventions: Other: Experimental formulas (EF)
- Control formulas (CF) group (Active Comparator): Starter infant formula, follow-up infant formula and growing-up milk (partially hydrolyzed bovine whey protein) not supplemented
  Interventions: Other: Control formulas (CF)
- Breastfed (BF) group (Active Comparator): Breast milk
  Interventions: Other: Breast feeding (BF)

INTERVENTIONS:
Other: Experimental formulas (EF) — First age formula administered orally ad libitum until 6 months of age, switch to second age formula until 12 months and finally to growing-up milk from 12 to 15 months
  Arms: Experimental formulas (EF) group
Other: Control formulas (CF) — First age formula administered orally ad libitum until 6 months of age, switch to second age formula until 12 months and finally to growing-up milk from 12 to 15 months
  Arms: Control formulas (CF) group
Other: Breast feeding (BF) — Exclusive breast feeding up to 4 months
  Arms: Breastfed (BF) group

SUMMARY:
This is a randomized, controlled, multicenter, double-blind study of healthy term infants. The primary objective of the trial is to demonstrate the safety of a a starter infant formula supplemented with pre- and probiotic(s) by comparing the growth of infants randomized to the experimental formula versus the control formula from enrolment to 4 months of age.

DETAILED DESCRIPTION:
This is a randomized, controlled, multicenter, double-blind study of healthy term infants, consisting of two randomized formula-fed arms (control and experimental formulas) and a non-randomized breast-fed reference group.

The population under investigation are healthy infants aged ≤14 days at enrollment. The planned sample size for formula-fed infants is 236 (118 per study group). A non-randomized breastfed reference group of 90 healthy, term, exclusively breastfed infants up to 4 months will also be enrolled.

Study formulas are administrated orally, ad libitum, from enrollment until 15 months of age.

The primary objective of the trial is to demonstrate the safety of a starter infant formula supplemented with pre- and probiotic(s) by comparing the growth (weight gain, g/day) of infants randomized to the experimental formula versus the control formula from enrolment to 4 months of age.

In addition fecal microbiome, fecal metabolic profile, fecal markers of immune and gut health, blood markers of immune health (in a subset of 60 infants/group), GI tolerance, bone index (subset of 40 infants/group), other anthropometric measurements, dietary pattern and infant illness and infection outcomes will be assessed/measured.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the infant's parent(s)/ legally accepted representatives LAR have been informed of all pertinent aspects of the study.
2. Infants whose parent(s)/LAR have reached the legal age of majority in the countries where the study is conducted.
3. Infants whose parent(s)/LAR are willing and able to comply with scheduled visits, and the requirements of the study protocol.
4. Infants whose parent(s)/LAR are able to be contacted directly by telephone throughout the study.
5. Infants must meet all of the following inclusion criteria to be eligible for enrollment into the study:

   1. Healthy term infant (≥37 weeks of gestation)
   2. At enrollment visit, post-natal age ≤14 days/0.5 months
   3. Birth weight ≥ 2500g and ≤ 4500g.
   4. For formula-fed groups, infants must be exclusively consuming and tolerating a cow's milk infant formula at time of enrollment and their parent(s)/LAR must have independently elected, before enrollment, not to breastfeed.
   5. For the breastfed group, infants must have been exclusively consuming breast milk since birth, and their parent(s)/LAR must have made the decision to continue exclusively breastfeeding until at least 4 months of age.

Exclusion Criteria:

1. Infants with conditions requiring infant feedings other than those specified in the protocol.
2. Infants who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   1. Evidence of major congenital malformations (e.g., cleft palate, extremity malformation)
   2. Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis)
   3. Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the infant inappropriate for entry into the study. Of note, children who are normally healthy but at the time of enrollment suffering from acute illness in a minor condition which are common in childhood and do not require some of the exclusionary medication mentioned below can be enrolled.
3. Infants who are presently receiving or have received prior to enrollment any of the following: medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool microbiota and characteristics (e.g., oral or systemic antibiotics, glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g. insulin or growth hormone); gastric acid secretion.
4. Currently participating or having participated in another clinical trial since birth.
5. Subjects or subjects' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Weight | From baseline (≤14 days) to 4 months of age
  Weight gain measured as mean daily weight gain in g/day

SECONDARY OUTCOMES:
Bifidobacteria abundance | At 90 days (3 months of age)
  Bifidobacteria abundance
Fecal microbiome | Stool sample collected at ≤14 days (baseline), 3, 6, 12 and 15 months of age
  Overall fecal microbiota composition, diversity, different bacteria taxa and microbiota community types assessed using next generation sequencing (NGS) technology
Fecal metabolic profile: fecal pH | Stool sample collected at ≤14 days (baseline), 3, 6, 12 and 15 months of age
  Fecal pH
Fecal metabolic profile: fecal organic acids | Stool sample collected at ≤14 days (baseline), 3, 6, 12 and 15 months of age
  Fecal organic acids (such as, but not restricted to lactate, including indole-lactate, L- and D-lactate, propionate, butyrate, acetate, valerate, and total fecal organic acids)
Fecal markers of immune health and gut barrier | Stool sample collected at ≤14 days (baseline), 3, 6, 12 and 15 months of age
  Fecal markers of immune health and gut barrier such as total secretory IgA (sIgA), lipocalin-2, calprotectin, and α-1-antitrypsin assessed by ELISA.
Fecal cytokine profile | Stool sample collected at ≤14 days (baseline), 3, 6, 12 and 15 months of age
  Fecal cytokine profile (such as but not restricted to: IL-6, IL-8, IL-1b, IL-22, IFN-γ) using multiplex assays
Blood markers of immune health | At 4 months of age
  Vaccine specific antibodies assessed by ELISA and Immuno-phenotyping in a subset of 120 infants (60/group)
GI-related behavior: stool frequency | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Stool frequency recorded via the GI Symptom and Behavior Diary
GI-related behavior: stool consistency | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Stool consistency recorded via the GI Symptom and Behavior Diary
GI-related behavior: incidence of spitting | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Incidence of spitting recorded via the GI Symptom and Behavior Diary
GI-related behavior: incidence of flatulence | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Incidence of flatulence via the GI Symptom and Behavior Diary
GI-related behavior: crying time | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Crying time via the GI Symptom and Behavior Diary
GI-related behavior: sleep time | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Sleep time via the GI Symptom and Behavior Diary
GI-related behaviour: volume of formula consumed | Retrospective 1-day (at baseline) and prospective for 3 days prior to 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Volume of formula consumed at each feeding or the number of breast milk feedings recorded via the GI Symptom and Behavior Diary
Infant Gastrointestinal Symptom Index | At baseline, 1, 2, 3, 4, 6, 9, 12 and 15 months of infant age
  GI symptoms via the Infant Gastrointestinal Symptom Questionnaire (IGSQ-13)
Bone index | At baseline, 3, 6, 9, 12 and 15 months of infant age
  Bone index measurement will be conducted using a non-invasive and radiation-free ultra-sound sonometer in a subset of 80 children (40/group)
Additional growth parameters: weight | At infant age ≤14 days (baseline), 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Weight in grams and corresponding weight-for-age Z-score according WHO growth standards
Additional growth parameters: length | At infant age ≤14 days (baseline), 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Length in centimeters and corresponding length-for-age Z-score according WHO growth standards
Additional growth parameters:head circumference | At infant age ≤14 days (baseline), 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  Head circumference in centimeters and corresponding head circumference-for-age Z-score according WHO growth standards
Additional growth parameters: Body Mass Index | At infant age ≤14 days (baseline), 1, 2, 3, 4, 6, 9, 12 and 15 months of age
  BMI (kg/m2) and corresponding BMI-for-age Z-score according WHO growth standards
Dietary pattern | At infant age 6, 9, 12 and 15 months
  Data collected using a food frequency questionnaire including key food groups for infants and young children
Absenteeism (infant and parent) | Data collected continuously from enrollment until 15 months of age
  Time away from daycare (infant) or work (parent) will be recorded during occurrences of illness / infection using a calendar-based electronic Infant Illness Diary (IID)

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (5):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Kinderartsen Huis, Hasselt
  - CHC-Groupe santé, Clinique MontLégia, Liège
  - CHU de Liège - CHR de la Citadelle, Liège
- France (6):
  - CHU Amiens-Picardie, Amiens
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital de la Croix Rousse, Lyon
  - CHU de Nantes, Nantes
  - CHU Charles Nicolle, Rouen
  - Hôpital Bretonneau, CHRU de Tours, Tours
- Germany (2):
  - Klinikum Südstadt Rostock, Rostock
  - Evangelisches Waldkrankenhaus Spandau, Spandau
- Spain (5):
  - Hospital Vithas Castellón, Castellon
  - Reina Sofía University Hospital, Córdoba
  - Instituto Hispalense de Pediatría, Unidad de Investigación, Seville
  - Hospital Vithas Valencia, Valencia
  - Quironsalud Valencia Hospital, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Picaud JC, Claris O, Gil-Campos M, De La Cueva IS, Cornette L, Alliet P, Leke A, Castanet M, Piloquet H, de Halleux V, Mitanchez D, Vandenplas Y, Maton P, Jochum F, Olbertz D, Policarpo SN, Lavalle L, Fumero C, Rodriguez-Garcia P, Moll JM, Silva-Zolezzi I, Zemrani B, Hays NP, Sprenger N, Miranda-Mallea J. Partially hydrolyzed, whey-based infant formula with six human milk oligosaccharides, B. infantis LMG11588, and B. lactis CNCM I-3446 is safe, well tolerated, and improves gut health: a staged analysis of a randomized trial. Front Nutr. 2025 Jul 23;12:1628847. doi: 10.3389/fnut.2025.1628847. eCollection 2025. PMID 40771223